CLINICAL TRIAL: NCT03892369
Title: Physiological Effects of FGF21 in Humans and Its Pathophysiological Role in Alcohol Dependence
Brief Title: FGF21 and Its Role in Alcohol Dependence
Acronym: AlcoDep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Head of Clinical Metabolic Physiology, Principal Investigator, Clinical Professor, PhD, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-18063495
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Abuse or Dependence
Keywords: Alcohol; FGF21; Alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Three matched groups. Group A: participants diagnosed with alcohol dependence, group B: participants with a father diagnosed with alcohol dependence, and C: a healthy control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol (Experimental): The participant receive 0.5 g ethanol per kg body weight over 10 minutes. Subsequently blood samples are taken frequently the next ten hours.
  Interventions: Other: Ethanol

INTERVENTIONS:
Other: Ethanol — Ethanol administration

SUMMARY:
Plasma fibroblast growthfactor-21 (FGF21) responses to acute alcohol exposure will be evaluated in three groups: A: 15 individuals diagnosed with alcohol dependence (ICD10 code F10.2) and no alcoholic liver diseases, B: 15 healthy individuals with one or two parents with alcohol dependence, and C: 15 healthy matched controls without history of or disposition to alcohol dependence. The experimental day consists of a load of 0.5 g ethanol per kg body weight ingested from time 0-10 minutes followed by a 7 h period in which blood will be sampled with frequent intervals, rating of preference for ethanol, salt, sour, bitterly and sweets, sensations of hunger, appetite, satiety, headache, and nausea will be evaluated using visuel analogue scale and resting energy expenditure will be evaluated using indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Caucasian males between 25 and 65 years of age
* BMI between 19 and 27 kg/m2
* Normal haemoglobin
* Normal fasting plasma glucose concentration (< 6 mmol/l) and normal glycated haemoglobin A1c (HbA1c) (< 42 mmol/mol)

Participants with a father diagnosed with alcohol dependence (group B):

* Father diagnosed with alcohol dependence
* Weekly alcohol intake of less than 14 units of alcohol (of 12 g)
* Normal Alcohol Use Disorders Identification Test (AUDIT) score

Healthy participants (group C):

* Weekly alcohol intake of less than 14 units of alcohol (of 12 g)
* Normal AUDIT score

Exclusion Criteria:

* Liver disease evaluated by plasma alanine aminotransferase (ALAT) > 3 × normal level, an international normalised ratio (INR) below normal values, or biopsy-verified alcoholic liver disease
* Diabetes mellitus
* Anaemia
* Nephropathy
* Other diseases the investigator finds disruptive for participation in the study.

Participants with a father diagnosed with alcohol dependence (group B):

- Former alcohol dependence or abuse

Healthy participants (group C):

* First-degree relatives with diabetes, liver disease and/or alcohol dependence
* Former alcohol dependence

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Fibroblast growthfactor-21 | One year
  Plasma FGF21 concentrations, a member of the endocrine FGF-family

SECONDARY OUTCOMES:
Ethanol | One year
  Plasma ethanol concentration
Glucose | One year
  Plasma glucose concentrations
Insulin and C-peptide | One year
  Serum insulin and C-peptide concentrations
Glucagon | One year
  Plasma glucagon concentration
Tumor Necrosis Factor-alpha (TNF) | One year
  Plasma TNF-alpha concentrations
Lipopolysaccharide Binding Protein (LBP) | One year
  Plasma LBP concentrations
Interferon-gamma (INF) | One year
  Plasma INF-gamma concentrations
Interleukine-10 (IL-10) | One year
  Plasma IL-10 concentrations
Interleukine-8 (IL-8) | One year
  Plasma IL-8 concentrations
Interleukine-6 (IL-6) | One year
  Plasma IL-6 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, Principal Investigator — Clinical Metabolic Physiology, Steno Diabetes Center Copenhagen
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark